CLINICAL TRIAL: NCT01371825
Title: An Open Label, Multicenter, Dose Escalation Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of SBC-102 (Sebelipase Alfa) in Children With Growth Failure Due to Lysosomal Acid Lipase Deficiency
Brief Title: Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of Sebelipase Alfa in Children With Growth Failure Due to Lysosomal Acid Lipase Deficiency
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL-CL03; NCT01473875 (obsolete NCT alias)
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Lysosomal Acid Lipase Deficiency; Wolman Disease
Keywords: LIPA; Wolman Disease; Wolman Phenotype; Acid Lipase Deficiency; Acid Cholesteryl Hydrolase; Acid Lipase Disease Deficiency, type 2; Cholesteryl Ester Storage Disease (CESD); Cholesteryl Ester Hydrolase Deficiency; Early Onset Lysosomal Acid Lipase Deficiency (Wolman Disease); LAL Deficiency; Late Onset Lysosomal Acid Lipase Deficiency (CESD); Wolman Disease (early onset LAL Deficiency); Related Disorders:; Non-alcoholic Fatty Liver Disease (NAFLD); Non-alcoholic Steatohepatitis (NASH); Alcoholic Liver Disease; Cryptogenic Cirrhosis; Niemann-Pick Disease (NPD) Type C; Chanarin Dorfman Syndrome
MeSH Terms: conditions — Wolman Disease; Cholesterol Ester Storage Disease; Non-alcoholic Fatty Liver Disease; Liver Diseases, Alcoholic; Cirrhosis, Cryptogenic; Niemann-Pick Diseases; Chanarin-Dorfman Syndrome | interventions — Sebelipase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-Label Sebelipase Alfa (Experimental): Participants received intravenous (IV) infusions of sebelipase alfa during the open-label treatment. Participants initially received 0.35 milligrams (mg)/kilogram (kg) qw and escalated to 1 mg/kg qw after demonstrating acceptable safety and tolerability during at least 2 infusions. One participant initiated treatment under a Temporary Use Authorization prior to enrollment, wherein the participant's dose was gradually escalated from 0.2 to 1 mg/kg over 4 weeks; the participant started the study at this dose. Participants on treatment for 96 weeks and on stable qw dosing for 24 weeks could be switched to an every other week (qow) dosing schedule. In the event of protocol-defined disease progression at any time during treatment, a participant could receive a dose increase from 1 to 3 mg/kg qw and, if necessary, a dose increase to 5 mg/kg qw with Safety Committee approval. Participants dosed qow who met dose-escalation criteria were reverted to qw dosing or escalated to 1 or 3 mg/kg qow.
  Interventions: Drug: Sebelipase alfa (SBC-102)

INTERVENTIONS:
Drug: Sebelipase alfa (SBC-102) — Sebelipase alfa is a recombinant human lysosomal acid lipase enzyme. The investigational medicinal product is an enzyme replacement therapy intended for treatment of participants with LAL Deficiency. Dosing occurred qw for up to 5 years.

SUMMARY:
This was an open-label, repeat-dose, intra-participant dose-escalation study of SBC-102 (sebelipase alfa) in children with growth failure due to lysosomal acid lipase (LAL) Deficiency. Eligible participants received once-weekly (qw) infusions of sebelipase alfa for up to 5 years.

DETAILED DESCRIPTION:
LAL Deficiency is a rare autosomal-recessive lipid storage disorder that is caused by a marked decrease or almost complete absence of LAL, leading to the accumulation of lipids, predominately cholesteryl esters and triglycerides, in various tissues and cell types. In the liver, accumulation of lipids leads to hepatomegaly, liver dysfunction, and hepatic failure. Although a single disease, LAL Deficiency presents as a clinical continuum with 2 major phenotypes, Cholesteryl Ester Storage Disease (CESD) and Wolman Disease.

Early-onset LAL Deficiency (Wolman Disease) is extremely rare, with an estimated incidence of less than 2 lives per million. It is characterized by profound malabsorption, growth failure, and hepatic failure, and is usually fatal in the first year of life.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent or legal guardian provided written informed consent/permission prior to any study procedures.
* Male or female child with documented decreased LAL activity relative to the normal range of the laboratory performing the assay or documented result of molecular genetic testing (2 mutations) confirming a diagnosis.
* Growth failure with onset before 6 months of age.

Exclusion Criteria:

* Clinically important concurrent disease or comorbidities.
* Had received an investigational product other than sebelipase alfa within 14 days prior to the first dose.
* Participant was older than 24 months of age.
* Myeloablative preparation, or other systemic pre-transplant conditioning, for hematopoietic stem cell or liver transplant.
* Previous hematopoietic stem cell or liver transplant.
* Known hypersensitivity to eggs.

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2011-05-04 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Irvine, California, United States
- Cairo, Egypt
- France (2):
  - Grenoble
  - Paris
- Dublin, Ireland
- United Kingdom (2):
  - London
  - Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jones SA, Rojas-Caro S, Quinn AG, Friedman M, Marulkar S, Ezgu F, Zaki O, Gargus JJ, Hughes J, Plantaz D, Vara R, Eckert S, Arnoux JB, Brassier A, Le Quan Sang KH, Valayannopoulos V. Survival in infants treated with sebelipase Alfa for lysosomal acid lipase deficiency: an open-label, multicenter, dose-escalation study. Orphanet J Rare Dis. 2017 Feb 8;12(1):25. doi: 10.1186/s13023-017-0587-3. PMID 28179030

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 centers participated in this study in the United Kingdom (UK), United States (US), France, Turkey, Ireland, and Egypt.
Pre-assignment Details: To assess eligibility, participants were screened for a period of up to 3 weeks prior to enrollment. 11 participants were screened, and 2 participants died during screening. The other 9 participants, all of whom were ≤8 months of age on the date of enrollment, met all eligibility criteria and were enrolled, treated, and analyzed.
Groups:
- Open-Label Sebelipase Alfa: Participants received intravenous (IV) infusions of sebelipase alfa during the open-label treatment. Participants initially received 0.35 milligrams (mg)/kilogram (kg) once weekly (qw) and escalated to 1 mg/kg qw after demonstrating acceptable safety and tolerability during at least 2 infusions. One participant initiated treatment under a Temporary Use Authorization prior to enrollment, wherein the participant's dose was gradually escalated from 0.2 to 1 mg/kg over 4 weeks; the participant started the study at this dose. Participants on treatment for 96 weeks and on stable qw dosing for 24 weeks could be switched to an every other week (qow) dosing schedule. In the event of protocol-defined disease progression at any time during treatment, a participant could receive a dose increase from 1 to 3 mg/kg qw and a dose increase to 5 mg/kg qw with Safety Committee approval. Participants dosed qow who met dose-escalation criteria were reverted to qw dosing or escalated to 1 or 3 mg/kg qow.
Period: Overall Study
Arm/Group | Open-Label Sebelipase Alfa
Started | 9
Received at Least 1 Dose of Study Drug | 9
Completed | 5
Not Completed | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Groups:
- Open-Label Sebelipase Alfa: Participants received IV infusions of sebelipase alfa during the open-label treatment. Participants initially received 0.35 mg/kg qw and escalated to 1 mg/kg qw after demonstrating acceptable safety and tolerability during at least 2 infusions. One participant initiated treatment under a Temporary Use Authorization prior to enrollment, wherein the participant's dose was gradually escalated from 0.2 to 1 mg/kg over 4 weeks; the participant started the study at this dose. Participants on treatment for 96 weeks and on stable qw dosing for 24 weeks could be switched to a qow dosing schedule. In the event of protocol-defined disease progression at any time during treatment, a participant could receive a dose increase from 1 to 3 mg/kg qw and, if necessary, a dose increase to 5 mg/kg qw with Safety Committee approval. Participants dosed qow who met dose-escalation criteria were reverted to qw dosing or escalated to 1 or 3 mg/kg qow.
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: months] | 3.41 [1.1 to 5.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants In The Primary Efficacy Analysis Set (PES) Surviving To 12 Months Of Age
Description: The primary efficacy endpoint was the percentage of participants (%) in the PES who survived to at least 12 months of age.
Time Frame: Month 12
Population: The PES included participants who received any amount of sebelipase alfa and who were ≤8 months of age on the date of their first infusion of sebelipase alfa. All 9 participants were included in the PES.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 9
Percentage of participants | 67 [29.9 to 92.5]

2. Secondary Outcome: Percentage Of Participants Surviving Beyond 12 Months Of Age
Description: The percentage of participants in the PES who survived to at least 18 months of age.
Time Frame: Baseline to Month 18, Month 24, Month 36, Month 48, and Month 60
Population: Evaluable participants in the PES, which included participants who received any amount of sebelipase alfa and who were ≤ 8 months of age on the date of their first infusion of sebelipase alfa. There were 2 non-evaluable participants at Month 60, defined as participants who were alive, still in the study, and had not yet reached 60 months of age.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 9
Percentage of participants
  Survival Through 18 Months of Age | 56 [21.2 to 86.3]
  Survival Through 24 Months of Age | 56 [21.2 to 86.3]
  Survival Through 36 Months of Age | 56 [21.2 to 86.3]
  Survival Through 48 Months of Age | 56 [21.2 to 86.3]
  Survival Through 60 Months of Age: number analyzed (Participants) | 7
  Survival Through 60 Months of Age | 43 [9.9 to 81.6]

3. Secondary Outcome: Median Age At Death
Description: Participants in the PES who died during the study, including 3 participants who died after having received between 1 and 4 infusions of sebelipase alfa and 1 participant who died after approximately 40 weeks on treatment.
Time Frame: Baseline to Week 260
Population: Participants in the PES who died during the study were included in this analysis. The PES included all 9 participants who received any amount of sebelipase alfa and who were ≤8 months of age on the date of their first infusion of sebelipase alfa.
Measure: Median (Full Range); unit: months
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 4
months | 3.63 [2.8 to 15.0]

4. Secondary Outcome: Change From Baseline To Months 12, 24, 36, 48, And 60 In Weight For Age (WFA) Percentiles
Description: Baseline is defined as the last measurement prior to the first infusion of sebelipase alfa.
Time Frame: Baseline, Month 12, Month 24, Month 36, Month 48, and Month 60
Population: as for outcome 1
Measure: Median (Full Range); unit: WFA Percentile
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 9
WFA Percentile
  Month 12: number analyzed (Participants) | 4
  Month 12 | 7.469 [5.35 to 13.77]
  Month 24: number analyzed (Participants) | 5
  Month 24 | 21.787 [0.91 to 30.37]
  Month 36: number analyzed (Participants) | 5
  Month 36 | 14.037 [-0.35 to 89.00]
  Month 48: number analyzed (Participants) | 5
  Month 48 | 15.770 [4.06 to 86.50]
  Month 60: number analyzed (Participants) | 5
  Month 60 | 19.869 [7.36 to 71.39]

5. Secondary Outcome: Number Of Participants With Stunting, Wasting, Or Underweight
Description: The number of participants who met criteria for the following dichotomous indicators of under nutrition were reported. These indicators included the following:
  * Stunting was defined as at least 2 standard deviations below the median for length-for-age/height-for-age;
  * Wasting was defined as wasting at least 2 standard deviations below the median for weight-for-length/weight-for-height; and
  * Underweight was defined as at least 2 standard deviations below the median for WFA.
Time Frame: Baseline to Month 12, Month 24, Month 36, Month 48, and Month 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 9
Participants
  Stunting, Baseline: number analyzed (Participants) | 8
  Stunting, Baseline | 4
  Stunting, Month 12: number analyzed (Participants) | 4
  Stunting, Month 12 | 1
  Stunting, Month 24: number analyzed (Participants) | 5
  Stunting, Month 24 | 0
  Stunting, Month 36: number analyzed (Participants) | 5
  Stunting, Month 36 | 0
  Stunting, Month 48: number analyzed (Participants) | 5
  Stunting, Month 48 | 0
  Stunting, Month 60: number analyzed (Participants) | 5
  Stunting, Month 60 | 0
  Wasting, Baseline: number analyzed (Participants) | 8
  Wasting, Baseline | 2
  Wasting, Month 12: number analyzed (Participants) | 4
  Wasting, Month 12 | 0
  Wasting, Month 24: number analyzed (Participants) | 5
  Wasting, Month 24 | 0
  Wasting, Month 36: number analyzed (Participants) | 5
  Wasting, Month 36 | 0
  Wasting, Month 48: number analyzed (Participants) | 5
  Wasting, Month 48 | 0
  Wasting, Month 60: number analyzed (Participants) | 5
  Wasting, Month 60 | 0
  Underweight, Baseline | 2
  Underweight, Month 12: number analyzed (Participants) | 4
  Underweight, Month 12 | 0
  Underweight, Month 24: number analyzed (Participants) | 5
  Underweight, Month 24 | 1
  Underweight, Month 36: number analyzed (Participants) | 5
  Underweight, Month 36 | 0
  Underweight, Month 48: number analyzed (Participants) | 5
  Underweight, Month 48 | 0
  Underweight, Month 60: number analyzed (Participants) | 5
  Underweight, Month 60 | 0
  No Stunting, Wasting, or Underweight, Baseline | 4
  No Stunting, Wasting, or Underweight, Month 12: number analyzed (Participants) | 4
  No Stunting, Wasting, or Underweight, Month 12 | 3
  No Stunting, Wasting, or Underweight, Month 24: number analyzed (Participants) | 5
  No Stunting, Wasting, or Underweight, Month 24 | 4
  No Stunting, Wasting, or Underweight, Month 36: number analyzed (Participants) | 5
  No Stunting, Wasting, or Underweight, Month 36 | 5
  No Stunting, Wasting, or Underweight, Month 48: number analyzed (Participants) | 5
  No Stunting, Wasting, or Underweight, Month 48 | 5
  No Stunting, Wasting, or Underweight, Month 60: number analyzed (Participants) | 5
  No Stunting, Wasting, or Underweight, Month 60 | 5

6. Secondary Outcome: Change From Baseline To Months 12, 24, 36, 48, And 60 In Serum Transaminases (ALT And AST)
Description: Change from Baseline to Months 12, 24, 36, 48, and 60 for alanine aminotransferase (ALT) and aspartate aminotransferase (AST).
Time Frame: Baseline, Month 12, Month 24, Month 36, Month 48, and Month 60
Population: as for outcome 1
Measure: Median (Full Range); unit: units/Liter (U/L)
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 9
units/Liter (U/L)
  ALT, Month 12: number analyzed (Participants) | 4
  ALT, Month 12 | -13.50 [-121.00 to 12.00]
  ALT, Month 24: number analyzed (Participants) | 5
  ALT, Month 24 | -5.00 [-111.00 to 228.00]
  ALT, Month 36: number analyzed (Participants) | 5
  ALT, Month 36 | -4.00 [-100.00 to 107.0]
  ALT, Month 48: number analyzed (Participants) | 4
  ALT, Month 48 | -27.50 [-129.00 to -2.00]
  ALT, Month 60: number analyzed (Participants) | 4
  ALT, Month 60 | -27.00 [-122.00 to 2.00]
  AST, Month 12: number analyzed (Participants) | 4
  AST, Month 12 | -43.50 [-62.00 to -29.00]
  AST, Month 24: number analyzed (Participants) | 5
  AST, Month 24 | -30.00 [-49.00 to 67.00]
  AST, Month 36: number analyzed (Participants) | 4
  AST, Month 36 | -33.00 [-49.00 to 86.00]
  AST, Month 48: number analyzed (Participants) | 5
  AST, Month 48 | -51.00 [-67.00 to -31.00]
  AST, Month 60: number analyzed (Participants) | 4
  AST, Month 60 | -40.00 [-84.00 to -17.00]

7. Secondary Outcome: Change From Baseline To Months 12, 24, 36, 48, And 60 In Serum Ferritin
Description: The median change in serum ferritin from Baseline to Months 12, 24, 36, 48, and 60 is presented.
Time Frame: Baseline, Month 12, Month 24, Month 36, Month 48, and Month 60
Population: as for outcome 1
Measure: Median (Full Range); unit: micrograms/Liter (µg/L)
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 9
micrograms/Liter (µg/L)
  Month 12: number analyzed (Participants) | 3
  Month 12 | -294.40 [-562.2 to -271.0]
  Month 24: number analyzed (Participants) | 3
  Month 24 | -239.00 [-298.0 to -235.0]
  Month 36: number analyzed (Participants) | 4
  Month 36 | -262.95 [-566.6 to -166.0]
  Month 48: number analyzed (Participants) | 3
  Month 48 | -268.00 [-278.0 to -179.0]
  Month 60: number analyzed (Participants) | 3
  Month 60 | -213.00 [-543.9 to -155.0]

8. Secondary Outcome: Number Of Participants Achieving And Maintaining Transfusion-free Hemoglobin Normalization [TFHN]
Description: The number of participants achieving and maintaining TFHN are presented.
  For TFHN to be achieved, the participant must a) have had 2 post-baseline measurements of hemoglobin at least 4 weeks apart that were both above the age-adjusted lower limit of normal; b) have had no known additional measurements of hemoglobin that were below the age-adjusted lower limit of normal during the (minimum) 4-week period; and c) have had no transfusions during the (minimum) 4-week period, and also no transfusions for 2 weeks prior to the first hemoglobin measurement in the (minimum) 4-week period.
  For TFHN to be maintained, the participant must have been transfusion-free beginning at Week 6 and had all hemoglobin assessments above the lower limit of normal beginning in Week 8 and lasting at least 13 weeks.
Time Frame: Baseline to Month 60
Population: Participants in the PES who received treatment with sebelipase alfa for at least 4 weeks (and could therefore be assessed for short-term TFHN). The PES included participants who received any amount of sebelipase alfa and who were ≤ 8 months of age on the date of their first infusion of sebelipase alfa.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 9
Participants
  Achieved TFHN | 6
  Maintained TFHN | 2

ADVERSE EVENTS:
Time Frame: Week 260
Description: Adverse events were obtained through spontaneous reporting or were elicited by specific questioning of the participant's parent or legal guardian. Treatment-emergent adverse events included events with an onset at or following the start of treatment with study drug or that worsened in severity or relationship at or following the start of treatment, and occurring up to 30 days after the last infusion of sebelipase alfa.
Arm/Group | Open-Label Sebelipase Alfa
All-Cause Mortality (participants affected / at risk) | 4/9
Serious Adverse Events (participants affected / at risk) | 9/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Sebelipase Alfa (N=9)
Pallor (Vascular disorders) | 1
Chills (General disorders) | 1
Pyrexia (General disorders) | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Hyperthermia (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Bacterial pyelonephritis (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 2
Device related infection (Infections and infestations) | 2
Device related sepsis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Roseola (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Weight decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Food intolerance (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Poor venous access (Vascular disorders) | 1
Tachycardia (Cardiac disorders) | 1
Sudden cardiac death (General disorders) | 1
Malabsorption (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Adenovirus infection (Infections and infestations) | 1
Amoebic dysentery (Infections and infestations) | 1
Croup infectious (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Rotavirus infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Open-Label Sebelipase Alfa (N=9)
Anaemia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 2
Cardiovascular disorder (Cardiac disorders) | 1
Hydrocele (Congenital, familial and genetic disorders) | 2
Ear pain (Ear and labyrinth disorders) | 2
Middle ear inflammation (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Conjunctivitis (Eye disorders) | 1
Pupillary disorder (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 6
Abdominal distension (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Teething (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Faeces discoloured (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 2
Post-tussive vomiting (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Tongue dicolouration (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 5
Chills (General disorders) | 1
Hyperthermia (General disorders) | 1
Catheter site rash (General disorders) | 1
Device dislocation (Product Issues) | 1
Disease progression (General disorders) | 1
Infusion Site Extravasation (General disorders) | 1
Feeling abnormal (General disorders) | 1
Gait disturbance (General disorders) | 1
Granuloma (General disorders) | 1
Infusion site oedema (General disorders) | 1
Irritability (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Rhinitis (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 5
Device related infection (Infections and infestations) | 2
Ear infection viral (Infections and infestations) | 2
Bronchiolitis (Infections and infestations) | 2
Catheter site infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 3
Varicella (Infections and infestations) | 3
Bacterial infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Candida nappy rash (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Eyelid infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Metapneumovirus infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral fungal infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Staphylococcal skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 3
Contusion (Injury, poisoning and procedural complications) | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Mouth injury (Injury, poisoning and procedural complications) | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Staphylococcus test positive (Investigations) | 1
Blood immunoglobulin A abnormal (Investigations) | 1
Blood immunoglobulin G abnormal (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood urea increased (Investigations) | 1
Body temperature increased (Investigations) | 1
Neutrophil count increased (Investigations) | 1
Norovirus test positive (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Platelet count increased (Investigations) | 1
Respiratory syncytial virus test positive (Investigations) | 1
Serum ferritin increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Urine albumin/creatinine ratio increased (Investigations) | 1
Urine output decreased (Investigations) | 1
Vitamin D decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 3
Hypotonia (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Penile blister (Reproductive system and breast disorders) | 1/5 — The AE of penile blister can only affect males, and there are 5 total males exposed.
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3
Eczema (Skin and subcutaneous tissue disorders) | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Umbilical erythema (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Pallor (Vascular disorders) | 1
Lymphocyte count increased (Investigations) | 1
Asthenia (General disorders) | 1
Catheter site pain (General disorders) | 1
Catheter site swelling (General disorders) | 1
Swelling (General disorders) | 1
Irritability (Psychiatric disorders) | 1
Emotional disorder (Psychiatric disorders) | 1
Genital rash (Reproductive system and breast disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Stoma site inflammation (Injury, poisoning and procedural complications) | 1
Tooth injury (Injury, poisoning and procedural complications) | 1
Lymphocyte count abnormal (Investigations) | 1
Monocyte count increased (Investigations) | 1
Adenovirus test positive (Investigations) | 1
Blood immunoglobulin G decreased (Investigations) | 1
Blood albumin decreased (Investigations) | 2
Clostridium test positive (Investigations) | 1
Parasite stool test positive (Investigations) | 1
Pseudomonas test positive (Investigations) | 1
Respirovirus test positive (Investigations) | 1
Vitamin E decreased (Investigations) | 1
Protein total decreased (Investigations) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Headache (Nervous system disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Xanthoma (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Device malfunction (Product Issues) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Vitamin A deficiency (Metabolism and nutrition disorders) | 1
Vitamin E deficiency (Metabolism and nutrition disorders) | 2
Vitamin K deficiency (Metabolism and nutrition disorders) | 2
Angular cheilitis (Infections and infestations) | 1
Croup infectious (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Infectious mononucleosis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Scarlet fever (Infections and infestations) | 1
Stoma site candida (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 2
Hand-foot-and-mouth disease (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Ear infection (Infections and infestations) | 3
Conjunctivitis (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-01-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT01371825/Prot_000.pdf
  • Statistical Analysis Plan (2014-03-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT01371825/SAP_001.pdf